CLINICAL TRIAL: NCT04112199
Title: A Phase 2 Randomized, Dose-Titration, Open-Label Study Evaluating the Safety and Efficacy of BIV201 Compared to Standard of Care to Reduce Ascites and Complications in Cirrhotic Patients With Refractory Ascites
Brief Title: A Study for Evaluation of BIV201 to Reduce Ascites and Complications in Patients With Cirrhosis and Refractory Ascites
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: For reasons unrelated to safety or efficacy
Sponsor: BioVie Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIT-002
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Ascites; Decompensated Cirrhosis
Keywords: Terlipressin; Refractory ascites
MeSH Terms: conditions — Ascites

STUDY DESIGN:
Intervention Model Description: Thirty patients will be randomized to either BIV201 continuous infusion plus SOC or SOC alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIV201 plus Standard of Care (Experimental): BIV201 continuous infusion - treatment for two 28 day cycles.
  Interventions: Drug: BIV201 continuous infusion
- Standard of care (No Intervention): Per AASLD guidelines: diuretics and therapeutic paracentesis

INTERVENTIONS:
Drug: BIV201 continuous infusion — BIV201 continuous infusion with terlipressin for a total of two 28 day cycles. Initiate treatment at 3 mg per 24 hour period and titrate stepwise up to a maximum of 8 mg per 24 hour period based on tolerability and response.
  Other Names: terlipressin diacetate
  Arms: BIV201 plus Standard of Care

SUMMARY:
This study evaluates the addition of BIV201 (terlipressin diacetate) as a continuous infusion in addition to standard of care (diuretics and therapeutic paracentesis) for reduction of ascites and complications in adult patients with refractory ascites secondary to decompensated cirrhosis

DETAILED DESCRIPTION:
Terlipressin has been shown to reduce portal hypertension, improve renal function and induce natriuresis in cirrhotic patients with ascites without hepatorenal syndrome (HRS). It is approved in Europe for the treatment of bleeding esophageal varices and HRS type 1 and is usually administered as an IV bolus starting at 1 mg every 6 h and increased to 2 mg every 6 h (maximum 8 mg/day depending on response).

This study will evaluate the use of terlipressin delivered by continuous infusion for two 28 day treatment cycles for reduction of ascites accumulation and complications in adult patients with refractory ascites secondary to decompensated cirrhosis. Continuous infusion allows for a significant reduction in the daily effective dose required for treatment and improved safety of terlipressin delivered as a low-dose continuous infusion could enable its use in the outpatient setting in the prolonged treatment of patients with refractory ascites.

ELIGIBILITY:
Inclusion Criteria

* Informed consent prior to any study-related procedures
* Male or female patients age 18 to 75 years old
* Cirrhosis of the liver (Non-alcoholic steatohepatitis, alcohol, viral and autoimmune)
* Patient has diuretic-resistant, intractable ascites or is unsuitable for treatment with diuretics and required:

  o In the 60-day period from the last LVP before consent, required, between 3 and 9 LVPs, including the last LVP on or before the day of consent.
* Dates for all LVPs that occurred within 90 days prior to consent have been recorded. The volume of ascites removed at each of the LVPs must also have been recorded for the 90-day period prior to the last LVPs before consent
* Serum creatinine (SCr) ≤2.00 mg/dL determined prior to randomization
* Women of child-bearing potential (e.g. not post-menopausal for at least one year or surgically sterile) must be neither pregnant nor lactating and must agree to use adequate birth control or be abstinent for the duration of the study
* If patient is treated with ACE inhibitors or beta blockers, dose has been stable for at least 30 days prior to randomization and may be maintained on that dose for the trial duration
* If patient is treated with diuretics, patient has been on a stable daily dose for at least 10 days prior to consent
* Willing and able to comply with trial instructions

Exclusion Criteria

* Ascites with causes other than cirrhosis; such as cardiac or nephrogenic ascites or malignant ascites due to peritoneal carcinomatosis
* Urinary sodium excretion >100 mmol/day between day of consent and randomization
* Total bilirubin >5 mg/dL
* Blood clotting International normalized ratio (INR) >2.5
* Current or recent (within 3 months of consent) renal replacement therapy
* Current or recent (within 3 month of consent) hepatic encephalopathy Grade 3 or 4 (West-Haven)
* Superimposed acute liver failure/injury due to factors including acute alcoholic hepatitis, acute viral hepatitis, drugs, medications (e.g., acetaminophen), or other toxins (e.g., mushroom [Amanita] poisoning)
* History or presence of hepatic hydrothorax, known pulmonary hypertension and a history of hepatopulmonary syndrome
* Current or recent treatment (within 7 days of randomization) with octreotide, midodrine, vasopressin, dopamine or other vasopressors
* Current or recent (in the previous 60 days from consent) episode of respiratory failure requiring positive airway pressure (PAP) devices or intubation
* Sepsis episode in the previous 28 days from consent
* Episode of SBP within the 28 days prior to consent
* Episode of gastrointestinal hemorrhage (non-variceal) within 28 days prior to consent
* Episode of esophageal variceal bleed within one week prior to consent
* Ongoing documented or suspected infection
* Severe cardiovascular disease that is a contraindication to terlipressin therapy such as a history of myocardial infarction, angina pectoris, advanced arteriosclerosis, uncontrolled cardiac arrhythmia, severe coronary insufficiency or uncontrolled hypertension
* Findings suggestive of severe organic renal disease (severe proteinuria/hematuria, or abnormal renal ultrasound suggestive of obstructive renal pathology)
* Use of nephrotoxic drugs (e.g., aminoglycosides) in the 4 weeks before screening
* Severe comorbidity that in the opinion of the Investigator would affect short-term prognosis and/or disallow safe participation in the trial (such as for example, severe anemia or pancytopenia, advanced progressive neoplasia such as hepatocellular carcinoma, unless eligible for transplant)
* Patient who, in the judgment of the investigator, has been an excessive alcohol drinker in the past 12 weeks
* Patient is in the opinion of the investigator, despite previous education on sodium restriction, anticipated to remain grossly non-compliant of sodium restricted diet
* Implanted alfapump or previous recipient of alfapump that had pump removed within past 3 months
* Recipient of renal or liver transplant
* Planned elective surgery related to cirrhosis complications, for example for hernia repair
* Known allergy or hypersensitivity to terlipressin
* Participation in other clinical research studies involving the treatment with other investigational drugs or evaluation with implantable devices within 30 days of consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-17 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
Incidence of complications, at least grade 2 severity | 180 days following randomization
  Incidence of complications, at least grade 2, during the 180 days following randomization

SECONDARY OUTCOMES:
Change in cumulative ascites | 12 weeks
  Change in cumulative ascites during the first 12 weeks following randomization versus the 12 weeks pre-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Palumbo, MD, Study Director — BioVie Inc.
Locations (10):
- United States (10):
  - UCLA, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Mercy Medical Center, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for primary and secondary end-points may be made available after NDA filing.